CLINICAL TRIAL: NCT02157311
Title: Evaluation of the Capacity of a Weekly Strategy of 4 Consecutive Days on Treatment Followed by 3 Days Off Treatment, in HIV-1 Infected Patients With Undetectable Viral Load for at Least 12 Months, to Maintain a Virological Success With This Intermittent Maintenance Therapy After a Successful Continuous Induction Therapy.
Brief Title: 4 Consecutive Days on Treatment Followed by 3 Days Off Treatment, in HIV Patients
Acronym: ANRS162-4D
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ANRS162-4D; 2014-000146-29 (EudraCT Number)
Record Dates: First submitted 2014-05-21; First posted 2014-06-06 (Estimated); Last update posted 2016-01-27 (Estimated); Status verified 2016-01

CONDITIONS: HIV-1 Infection
Keywords: HIV-1; simplification,; treatment discontinuation; virological success; four days a week
MeSH Terms: interventions — Tenofovir; Emtricitabine; abacavir; Lamivudine; efavirenz; Rilpivirine; etravirine; atazanavir, ritonavir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Four consecutive days on treatment and 3 days off (Experimental): All patients will take a combination of three HIV treatment with a weekly strategy of 4 consecutive days on treatment followed by 3 days off treatment
  Interventions: Drug: Four consecutive days on treatment and 3 days off

INTERVENTIONS:
Drug: Four consecutive days on treatment and 3 days off — All patients will take a combination of three of these treatment with a weekly strategy of 4 consecutive days on treatment followed by 3 days off treatment
  Other Names: tenofovir,; emtricitabine,; abacavir,; lamivudine,; efavirenz,; rilpivirine,; etravirine,; lopinavir/r,; darunavir/r,; atazanavir/r

SUMMARY:
Evaluate after 48 weeks, the capacity of a weekly strategy of 4 consecutive days on treatment followed by 3 days off treatment, in HIV-1 treated patients with undetectable viral load for at least 12 months and continuous antiretroviral regimen unchanged for at least 4 months, to maintain a therapeutic success defined by the absence of virological failure (2 consecutive viral loads > 50 cp/mL) and the absence of interruption of therapeutic strategy (interruption or change of the " 4 days on / 3 days off " strategy for a time longer than 30 consecutive days).

DETAILED DESCRIPTION:
Methods:

Open-label, multicentric, prospective, non-randomized, non-controlled trial to evaluate at 48 weeks, the capacity of a weekly strategy of 4 consecutive days on treatment followed by 3 days off treatment, in HIV-1 treated patients with undetectable viral load for at least 12 months and continuous antiretroviral regimen unchanged for at least 4 months, to maintain a therapeutic success defined by the absence of virological failure (2 consecutive viral loads > 50 cp/mL) and the absence of interruption of therapeutic strategy (interruption or change of the " 4 days on / 3 days off " strategy for a time longer than 30 consecutive days).

Allocation: Non-randomized Endpoint Classification: Safety/Efficacy Study Primary Purpose: Treatment

Enrollment: 100 patients

ELIGIBILITY:
Inclusion Criteria:

* • HIV-1 documented infection

  * Age 18 years or older
  * HIV-1 viral load always ≤ 50 cp/mL for at least 12 months (with a minimum of 3 measures in the last 12 months, including screening)
  * CD4+ lymphocytes count > 250/mm3, for at least 6 months
  * Treatment with a stable regimen for at least 4 months prior to screening, containing 2 nucleoside/nucleotide analog reverse transcriptase inhibitors (NRTI) combined with, either 1 non-nucleoside reverse transcriptase inhibitor (NNRTI), or 1 ritonavir-boosted protease inhibitor (PI/r). The list of accepted antiretroviral drugs is limited to :

    1. NRTI : tenofovir, emtricitabine, abacavir, lamivudine
    2. PI/r : lopinavir/r, darunavir/r or atazanavir/r
    3. NNRTI : efavirenz, rilpivirine or etravirine.
  * Exclusive antiretroviral 3 drug-therapy (no 4 drug-therapy)
  * A least one genotypic resistance test available (reverse transcriptase and/or protease amino acid sequence, according to on-going antiretroviral drugs) ; on each genotypic resistance test(s) available in medical history, susceptibility to every on-going antiretroviral drugs must be demonstrated
  * Clearance of the creatinine > 60 mL/min (MDRD)
  * ASAT and ALAT < 3 ULN
  * Hemoglobin > 10 g/dl
  * Platelets count > 100 000/mm3
  * Negative pregnancy test for potential child-bearing women and mechanical contraception for sexual intercourses
  * Patient living in France and affiliated to a social security system
  * Written informed consent

Exclusion Criteria:

* • HIV-2 infection

  * HBV infection (positive HBs antigen) or isolated positive HBc antibody
  * HCV infection requiring specific treatment during the 51 weeks of the trial
  * At least one known resistance to one of on-going antiretroviral drugs
  * Exclusive antiretroviral 3 drug-therapy (no 4 drug-therapy)
  * No genotypic resistance test available
  * On-going either interferon, interleukin treatment, or every immuno- / chemo-therapy
  * Progressive opportunistic infection, on-going treatment for opportunistic infection or tuberculosis
  * Patient with irregular follow-up or with treatment adherence problems
  * Any condition (alcohol, drug abuse…) compromising treatment adherence, treatment safety, and/or study adherence
  * Progressive neurological disorders (meningitis, encephalitis, myelitis…) related to HIV infection or not
  * Medical history of severe neuropsychiatric disorder, with insufficient treatment efficacy
  * Subject under legal guardianship or incapacitation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-07; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Capacity to maintain a therapeutic success with 4 days on treatment followed 3 days off treatment | Week 48
  To evaluate after 48 weeks, the capacity of a weekly strategy of 4 consecutive days on treatment followed by 3 days off treatment, in HIV-1 treated patients with undetectable viral load for at least 12 months and continuous antiretroviral regimen unchanged for at least 4 months, to maintain a therapeutic success defined by the absence of virological failure (2 consecutive viral loads > 50 cp/mL) and the absence of interruption of therapeutic strategy (interruption or change of the " 4 days on / 3 days off " strategy for a time longer than 30 consecutive days).

SECONDARY OUTCOMES:
Virological success | Week 48
  The HIV-1 viral load at week 48 must be inferior to 50 copies/mL
The time of virological failure occurrence | Week 0, Week 4, Week 8, Week 12, Week 16, Week 24, Week 32, Week 40, Week 48, Week 51
  Measure the delay between week 0 and the date of the different virologic failure
The blips | Week 0, Week 4, Week 8, Week 12, Week 16, Week 24, Week 32, Week 40, Week 48, Week 51
  Number of blips (viral load detectable on 1 sample) during the study
The low viral loads (between 20 - 50 cp/mL) | Week 0, Week 4, Week 8, Week 12, Week 16, Week 24, Week 32, Week 40, Week 48, Week 51
  Measurement of the low viral loads (between 20 - 50 cop/mL)
Detected signal on viral quantification | Week 0, Week 4, Week 8, Week 12, Week 16, Week 24, Week 32, Week 40, Week 48, Week 51
  The presence or not of detected signal when no quantification is possible on viral loads
Mutations resistance | Week 0, Week 4, Week 8, Week 12, Week 16, Week 24, Week 32, Week 40, Week 48, Week 51
  The profile of new resistance mutations in case of virological failure
Evaluation CD4, CD8 and CD4/CD8 ratios | Week 0, week 8, week 16, week 24, week 24, week 32, week 40 and week 48
  Measurement of the CD4 cell count, CD8 cell count, and CD4/CD8 ratio
HIV proviral DNA | Week 0, Week 24 and Week 48
  The evolution of HIV proviral DNA in the peripheral blood mononuclear cells (PBMC)
Clinical events related to HIV infection | Week 0, Week 4, Week 8, Week 12, Week 16, Week 24, Week 32, Week 40, Week 48, Week 51
  Clinical events related to HIV infection, according to the US CDC classification
Adverse events | Week 0, Week 4, Week 8, Week 12, Week 16, Week 24, Week 32, Week 40, Week 48, Week 51
  Collect all clinical and biological adverse events
Interruption or modification of the therapeutic strategy | Week 0, Week 4, Week 8, Week 12, Week 16, Week 24, Week 32, Week 40, Week 48, Week 51
  Every interruption or modification of the therapeutic strategy for more than 30 days
Renal parameters | Week 0, week 8, week 16, week 24, week 32, week 40 and week 48
  The evolution of creatinin and clearance of creatinin between week 0 and Week 48.
Inflammation and immune activation | Week 0, week 24 and Week 48
  The evolution of inflammation and immune activation parameters (IL-6, CRP-US, CD14s, IP-10 and MIG-1).
  The measurement will be done at the end of the study in a central lab on the biobank
Antiretrovirals Pharmacokinetic | Week 0, week 24 and week 48
  The evolution of pharmacokinetic parameters, for protease inhibitors (lopinavir, darunavir or atazanavir) or non-nucleoside reverse transcriptase inhibitors (efavirensz, etravirine or rilpivirine) The measurment will be done on the sample bank at the end of the study in a central lab
Antiretrovirals pharmacokinetic | week 4, week8, week 12, week 24, week 32 and week 48
  Measurment of Residual plasmatic concentrations of protease inhibitors (lopinavir/r - darunavir/r - atazanavir/r ) or non-nucleoside reverse transcriptase inhibitors (efavirenz or rilpivirine or etravirine), at the end of the 3-days off, from Day 0 to week 48.
  The measurment will be done on the sample bank at the end of the study in a central lab
Quality of life | week 0, week 24 and week 48
  selfquestionnary to measure the quality of life (PRO-QOL HIV and felt symptoms )
Adherence | Week 0, Week 4, Week 8, Week 12, Week 16, Week 24, Week 32, Week 40, Week 48, Week 51
  Measurement of treatment adherence (questionnaire, self-survey book, pharmacological measures of antiretroviral drugs, medication event monitoring system)
Hepatitis parameters | Week 0, week 8, week 16, week 24, week 32, week 40 and week 48
  Measurment of AST, SGOT, CGT
Glucidolipidics parameters | Week 0, week 24 and week 48
  Measurement of Glycemia, Triglycerids, total cholesterol, HDL and LDL

CONTACTS AND LOCATIONS:
Overall Officials: Christian PERRONNE, MD-PHD, Principal Investigator — Hôpital Raymond Poincaré; Jean-Claude MELCHIOR, MD-PHD, Principal Investigator — Hôpital Raymond Poincaré; Pierre DE TRUCHIS, MD, Principal Investigator — Hôpital Raymond Poincaré; Damien LE DU, MD, Principal Investigator — Hôpital Raymond Poincaré
Locations (17):
- France (17):
  - Hôpital Meynard, Fort-de-france, Martinique
  - Hôpital Avicenne, Bobigny
  - CHU Côte de Nacre, Caen
  - Centre Hospitalier Sud Francilien, Corbeil-Essonnes
  - Hôpital Le Bocage, Dijon
  - Hôpital Raymond Poincaré, Garches
  - Hôpital Bicêtre, Le Kremlin-Bicêtre
  - Hôpital Gui de Chauliac, Montpellier
  - Hôpital Saint-Antoine, Paris
  - Hôpital Pitié-Salpêtrière, Paris
  - Hôpital Européen Georges Pompidou, Paris
  - Hôpital Necker, Paris
  - Hôpital Bichat, Paris
  - Hôpital Tenon, Paris
  - Hôpital Foch, Suresnes
  - Hôpital Purpan, Toulouse
  - Hôpital Bretonneau, Tours

REFERENCES:
- [Derived] de Truchis P, Assoumou L, Landman R, Mathez D, Le Du D, Bellet J, Amat K, Katlama C, Gras G, Bouchaud O, Duracinsky M, Abe E, Alvarez JC, Izopet J, Saillard J, Melchior JC, Leibowitch J, Costagliola D, Girard PM, Perronne C; ANRS 162-4D Study Group. Four-days-a-week antiretroviral maintenance therapy in virologically controlled HIV-1-infected adults: the ANRS 162-4D trial. J Antimicrob Chemother. 2018 Mar 1;73(3):738-747. doi: 10.1093/jac/dkx434. PMID 29186458